CLINICAL TRIAL: NCT05981963
Title: A Phase 1, Single-center, Open-label Study to Evaluate the Pharmacokinetics, Metabolism, and Excretion of Orally Administered 60 mg BMS-986196, Including Radioactively Labeled [14C]-BMS-986196, in Healthy Male Participants
Brief Title: A Study to Evaluate the Drug Levels, Physical and Chemical Changes, and Removal of BMS-986196 in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IM038-1007
Record Dates: First submitted 2023-08-01; First posted 2023-08-08 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Healthy Male Volunteers
Keywords: Pharmacokinetics; BMS-986196; Healthy male volunteers; [14C]-BMS-986196; Total radioactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [14C]-BMS-986196 (Experimental)
  Interventions: Drug: [14C]-BMS-986196

INTERVENTIONS:
Drug: [14C]-BMS-986196 — Specified dose on specified days
  Other Names: BMS-986196

SUMMARY:
The purpose of this study is to evaluate the excretion pathway of orally administered [14C]-BMS-986196 and to assess the safety and tolerability of orally administered BMS-986196.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male participants without clinically significant deviation from normal in medical history, electrocardiogram (ECG), clinical laboratory determinations, and Day -1 physical examination.
* Body mass index of 18.0 to 35.0 kilograms/meter square (kg/m^2), inclusive, and total body weight ≥ 50 kg

Exclusion Criteria:

* Any significant acute or chronic medical illness as determined by the investigator.
* A history of clinically significant hepatic or pancreatic disease.
* Current or recent (within 3 months prior to study treatment administration) gastrointestinal disease that could impact upon the absorption, distribution, metabolism, or excretion of study treatment as determined by the investigator.

Note: Other protocol-defined inclusion/exclusion criteria apply.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2023-08-17 (Actual); Primary Completion 2023-10-22 (Actual); Study Completion 2023-10-22 (Actual)

PRIMARY OUTCOMES:
Total Radioactivity (TRA): Maximum observed plasma concentration (Cmax) | Up to Day 15
TRA: Time of Cmax (Tmax) | Up to Day 15
TRA: Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration (AUC [0-T]) | Up to Day 15
TRA: Amount of radioactivity recovered in urine (UR) | Up to Day 15
TRA: Amount of radioactivity recovered in feces (FR) | Up to Day 15
TRA: Amount of radioactivity recovered in bile (BR) | Up to 14 hours post dose
TRA: Percent of administered dose recovered in urine (%UR) | Up to Day 15
TRA: Percent of administered dose recovered in feces (%FR) | Up to Day 15
TRA: Total percent of administered dose recovered (urine, feces, and bile combined) (% Total) | Up to Day 15

SECONDARY OUTCOMES:
Cmax | Up to Day 15
Tmax | Up to Day 15
AUC (0-T) | Up to Day 15
Number of Participants with Adverse Events (AEs) | Up to Day 29
Number of Participants with Serious AEs (SAEs) | Up to Day 29
Number of Participants with AEs Leading to Discontinuation | Up to Day 29
Number of Participants with Vital Sign Abnormalities | Up to Day 15
Number of Participants with Electrocardiogram (ECG) Abnormalities | Up to Day 15
Number of Participants with Physical Examination Abnormalities | Up to Day 15
Number of Participants with Clinical Laboratory Abnormalities | Up to Day 15

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Labcorp Clinical Research Unit - Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSStudyConnect.com